CLINICAL TRIAL: NCT00078559
Title: The Use of Campath-1H, Tacrolimus, and Sirolimus Followed by Sirolimus Withdrawal in Renal Transplant Patients
Brief Title: Combination Immunosuppressive Therapy to Prevent Kidney Transplant Rejection in Adults
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: University of Wisconsin, Madison (Other)
Collaborators: Immune Tolerance Network (ITN) (Network)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: DAIT ITN013ST; H-2003-0435 (Other: HS IRB); NCT00585130 (obsolete NCT alias)
Record Dates: First submitted 2004-03-01; First posted 2004-03-02 (Estimated); Results first posted 2012-07-09 (Estimated); Last update posted 2018-06-29 (Actual); Status verified 2018-05

CONDITIONS: Kidney Transplantation; Kidney Disease
Keywords: Immunosuppression; Renal Failure
MeSH Terms: conditions — Kidney Diseases; Renal Insufficiency | interventions — Alemtuzumab; Sirolimus; Tacrolimus; Kidney Transplantation; Methylprednisolone; Acetaminophen; Diphenhydramine; Trimethoprim; Trimethoprim, Sulfamethoxazole Drug Combination; Acyclovir; Pentamidine; Clotrimazole; Nystatin

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Alemtuzumab (Experimental)
  Interventions: Drug: Alemtuzumab; Drug: Sirolimus; Drug: Tacrolimus; Procedure: Kidney transplant; Drug: Methylprednisolone (or equivalent); Drug: Acetaminophen; Drug: Diphenhydramine; Drug: Trimethoprim (TMP)/Sulfa (Bactrim, Septra); Drug: Valgancyclovir; Drug: Acyclovir; Drug: Pentamidine; Drug: Clotrimazole; Drug: Nystatin

INTERVENTIONS:
Drug: Alemtuzumab — 30mg intravenous infusion on days 0 (transplant), 1, and 2
Drug: Sirolimus — 2mg/day orally within 24-48 hrs post-transplant, and adjusted to achieve blood levels of 8-12 ng/mL for 1 year
Drug: Tacrolimus — 2mg orally twice daily, on days 1-60
Procedure: Kidney transplant — Kidney transplant with primary cadaveric or non-HLA-identical living donor kidney (0-3 HLA-antigen mismatch)
Drug: Methylprednisolone (or equivalent) — 250 mg intravenous infusion 60 minutes prior to first dose of alemtuzumab
Drug: Acetaminophen — 650 mg may be given 30-60 minutes prior to start of each infusion of alemtuzumab to prevent infusion related side effects such as fever, skin rash and pruritis
Drug: Diphenhydramine — 25 mg may be given 30-60 minutes prior to start of each infusion of alemtuzumab to prevent infusion related side effects such as fever, skin rash and pruritis
Drug: Trimethoprim (TMP)/Sulfa (Bactrim, Septra) — 1 double strength tablet 3 times a week from day 1 through 1 year post-transplant.
Drug: Valgancyclovir — Given orally beginning on day 1 for up to 10 days post-transplant (until participant discharged from hospital if prior to 10 days). Dose adjusted based on participants calculated creatinine clearance
Drug: Acyclovir — 400 mg orally twice daily or 800 mg orally four times daily (dose adjusted based on calculated creatinine clearance and cytomegalovirus antibody serologic status of donor and recipient) for a minimum of 3 months starting when valganciclovir discontinued.
Drug: Pentamidine — 300 mg/6 mL inhalation therapy once monthly for a total of 6 treatments. First treatment given within one week post-transplant for participants with a known allergy or intolerance to sulfa
Drug: Clotrimazole — 10 mg orally four times daily for a minimum of 3 months post-transplant (subjects take either clotrimazole or nystatin, not both)
Drug: Nystatin — 500,000 units/5 mL orally four times daily for a minimum of 3 months post-transplant (subjects take either nystatin or clotrimazole, not both)

SUMMARY:
Transplant rejection occurs when a patient's body does not recognize the new organ and attacks it. Patients who have kidney transplants must take drugs to prevent transplant rejection. Alemtuzumab is a man-made antibody used to treat certain blood disorders. The purpose of this study is to test the safety and effectiveness of using alemtuzumab in combination with two other drugs, sirolimus and tacrolimus, to prevent organ rejection after kidney transplantation. This study will also test whether this combination of medications will allow patients to eventually stop taking antirejection medications entirely.

Study hypothesis: A new strategy of immunosuppression using alemtuzumab, tacrolimus, and sirolimus for human renal transplantation will permit a step-wise withdrawal from immunosuppressive drugs.

DETAILED DESCRIPTION:
Drugs that suppress the immune system, such as sirolimus and tacrolimus, have contributed to increased success of transplantation. However, to prevent organ rejection, transplant recipients need to take immunosuppressive drugs for the rest of their lives, and these drugs make patients more susceptible to infection, endangering their health and survival. Regimens that are less toxic to or can eventually be withdrawn from transplant recipients are needed. Alemtuzumab is a monoclonal antibody that binds to and depletes excess T cells in the bone marrow of leukemia patients. This study will determine the effects of intravenous alemtuzumab and oral sirolimus and tacrolimus after kidney transplantation. The study will also evaluate this regimen's potential to allow eventual discontinuation of components of long-term immunosuppressive therapy.

This study will last up to 4 years. Participants will undergo kidney transplantation on Day 0 and will receive intravenous doses of alemtuzumab, acetaminophen, and diphenhydramine on Days 0, 1, and 2, as well as methylprednisolone on Day 0. After transplant, patients will receive up to 10 days of valganciclovir or acyclovir. Participants will take tacrolimus daily by mouth for at least 60 days after transplant and sirolimus daily by mouth for at least 12 months after transplant. As part of opportunistic infection (OI) prophylaxis, participants will also take sulfamethoxazole-trimethoprim by mouth 3 times a week, valganciclovir or acyclovir for up to 10 days post-transplant, and clotrimazole or nystatin by mouth for at least 3 months post-transplant.

There will be a minimum of 62 study visits spread out over 4 years after transplant. Vital signs measurement, adverse event and OI reporting, medication history, physical exam, and blood collection will occur at selected visits. Sirolimus withdrawal will begin when a participant meets certain study criteria. The withdrawal process will occur over a minimum of 3 months at an approximate rate of 33% of the pre-withdrawal dose per month. Participants eligible for sirolimus withdrawal will undergo several kidney biopsies, including one 2 weeks prior to the start of withdrawal, 6 and 12 months after completion of withdrawal, 1 year after study enrollment, and annually thereafter.

ELIGIBILITY:
Inclusion Criteria

* Kidney transplant with primary cadaveric or non-Human Leukocyte Antigen (HLA)-identical living donor kidney (0-3 HLA-antigen mismatch)
* Receiving only a kidney and no other organs
* Able to take medications by mouth
* Willing to use acceptable methods of contraception

Exclusion Criteria

* Received HLA-identical living-donor kidney transplant
* HLA-antigen mismatch greater than 3
* Panel reactive antibody (PRA) value greater than 10% at any time prior to enrollment
* Received a non-heart-beating donor allograft
* Received a kidney from a donor who is greater than 60 years of age
* End-stage Renal Disease (ESRD) due to Focal Segmental Glomulerosclerosis (FSGS)
* Previous kidney transplant
* Received multiorgan transplant
* Concomitant systemic corticosteroid therapy for other medical diseases
* Known hypersensitivity to alemtuzumab, tacrolimus, methylprednisolone, or sirolimus
* Human Immunodeficiency Virus (HIV) infected
* Hepatitis C virus infected
* Positive for hepatitis B surface antigen
* Received dual or en-bloc pediatric kidneys
* Anti-human Globulin (AHG) or T cell crossmatch positive
* Investigational drug within 6 weeks of study entry
* Known clinically significant cardiovascular or cerebrovascular disease
* Previous or current history of cancer or lymphoma. Patients with adequately treated basal or squamous cell skin carcinoma are not excluded.
* Clinically significant coagulopathy or a requirement for chronic anti-coagulation therapy precluding biopsy
* Cytomegalovirus (CMV)-negative recipient, if received kidney is from a CMV-positive donor
* History of a psychological illness or condition that, in the opinion of the investigator, may interfere with the study
* Graves disease. Patients who have been previously adequately treated with radioiodine ablative therapy are not excluded.
* Active systemic infections
* Platelets less than 100,000 cells/mm^3 at study entry
* Pregnant or breastfeeding

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 10 (Actual)
Dates: Start 2003-11; Primary Completion 2010-02 (Actual); Study Completion 2010-02 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: A. D'jamali, MD, MS, Principal Investigator — Immune Tolerance Network (ITN)
Locations (1):
- University of Wisconsin - Department of Medicine, Madison, Wisconsin, United States

REFERENCES:
- [Background] First MR. Tacrolimus based immunosuppression. J Nephrol. 2004 Nov-Dec;17 Suppl 8:S25-31. PMID 15599882
- [Background] Gourishankar S, Turner P, Halloran P. New developments in immunosuppressive therapy in renal transplantation. Expert Opin Biol Ther. 2002 Jun;2(5):483-501. doi: 10.1517/14712598.2.5.483. PMID 12079485
- [Background] Watson CJ, Bradley JA, Friend PJ, Firth J, Taylor CJ, Bradley JR, Smith KG, Thiru S, Jamieson NV, Hale G, Waldmann H, Calne R. Alemtuzumab (CAMPATH 1H) induction therapy in cadaveric kidney transplantation--efficacy and safety at five years. Am J Transplant. 2005 Jun;5(6):1347-53. doi: 10.1111/j.1600-6143.2005.00822.x. PMID 15888040
- See also: Click here for the Immune Tolerance Network Web site — http://www.immunetolerance.org
- See also: Related Info — http://www.niaid.nih.gov/

RESULTS

PARTICIPANT FLOW:
Recruitment Details: For this trial, one center in the United States enrolled ten eligible adult recipients of first kidney transplants (0-3 human leukocyte antigen (HLA)-antigen mismatch) from February 2005 to February 2006
Pre-assignment Details: At a screening visit, participants underwent procedures to establish inclusion/exclusion criteria and then sign the informed consent form. Refer to inclusion and exclusion criteria section for more details
Groups:
- Alemtuzumab: Recipients of first kidney transplants (0-3 HLA antigen mismatch) received induction therapy with alemtuzumab (1 dose [30 mg]each day, Days 0 [transplant day], 1 and 2, administered intravenously) , tacrolimus (the dose was initially 2 mg twice daily by mouth, and adjusted to maintain target blood levels of 4 to 8 ng/mL from Day 1 to Day 60) and sirolimus (the initial dose was 2 mg/day by mouth started <= 48 hours post-transplant, subsequently adjusted to achieve trough levels of 8 to 12 ng/mL through Month 12), followed by sirolimus withdrawal as tolerated
Period: Overall Study
Arm/Group | Alemtuzumab
Started | 10
Completed | 10 (1 subject stopped study drug due to a severe but non-serious AE, and completed the trial)
Not Completed | 0

BASELINE CHARACTERISTICS:
Arm/Group | Alemtuzumab
Number analyzed (Participants) | 10
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 10
  >=65 years | 0
Age, Continuous [Mean (Standard Deviation); unit: years] | 45.3 (10.5)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 3
  Male | 7
Region of Enrollment [Number; unit: participants]
  United States | 10
Primary Cause of Renal Failure [Number; unit: Participants]
  Glomerulonephritis | 0
  Pyelonephritis/Interstitial Nephritis | 0
  Cystic/Polycystic Kidney Disease | 4
  Hypertension | 0
  Diabetes Mellitus | 1
  Obstructive/Reflux Nephropathy | 1
  IgA Nephropathy | 2
  Post-streptococcal Glomerular Nephritis | 0
  Systemic Lupus Erythematosus | 0
  Etiology Uncertain | 2
  Other | 0
Pre-Transplant Dialysis [Number; unit: Participants] — Whether or not participant received dialysis pre-transplant and if they did, the type they received.
  Participants
    Hemodialysis and Peritoneal Dialysis | 0
    Hemodialysis | 5
    Peritoneal Dialysis | 0
    Dialysis - Unknown Type | 0
    Participants without pre-transplant dialysis | 5

OUTCOME MEASURES:

1. Primary Outcome: Number of Acute Rejections in All Enrolled Participants
Description: Number of acute rejections[1] in all enrolled subjects from the time of transplantation to the end of the trial (four years post-transplant)
  1. Acute rejection is defined as a biopsy-proven rejection: a renal biopsy demonstrates acute cellular or humoral rejection of Banff[2] Grade 1B or greater; or presumed rejection in the absence of biopsy-proven rejection, the participant is treated for an unexplained 20% increase in serum creatinine.
  2. Reference: Racusen LC, Solez K, Colvin RB et al,The Banff 97 working classification of renal allograft pathology. Kidney Int,55: 713-723, 1999
Time Frame: Four years post-transplant
Population: Intent-to-treat
Measure: Number; unit: Rejection Events
Arm/Group | Alemtuzumab
Number analyzed (Participants) | 10
Rejection Events | 1
Statistical Analysis 1: Comparison: Alemtuzumab; Test type: Superiority or Other; 95% Confidence Interval; Exact Binomial; Proportion with acute rejection = 0.1, 95% CI 2-sided [0.01 to 0.34]

2. Secondary Outcome: Number of Acute Rejections in All Enrolled Participants Following Sirolimus Withdrawal
Description: Following sirolimus withdrawal, the number of acute rejections[1] in all enrolled participants
  1] Acute rejection is defined as a biopsy-proven rejection: a renal biopsy demonstrates acute cellular or humoral rejection of Banff[2] Grade 1B or greater; or presumed rejection in the absence of biopsy-proven rejection, the participant is treated for an unexplained 20% increase in serum creatinine.
  [2] Reference: Racusen LC, Solez K, Colvin RB et al,The Banff 97 working classification of renal allograft pathology. Kidney Int,55: 713-723, 1999
Time Frame: Transplantation to end of study (up to four years post-transplant)
Population: Intent-to-treat
Measure: Number; unit: Rejection Events
Arm/Group | Alemtuzumab
Number analyzed (Participants) | 10
Rejection Events | 0
Statistical Analysis 1: Comparison: Alemtuzumab; Test type: Superiority or Other; 95% Confidence Interval; Exact Binomial; Proportion with acute rejection = 0, 95% CI 2-sided [0.0 to 0.3]

3. Secondary Outcome: Number of Acute Rejections Between Initiation of Sirolimus Withdrawal and End of Study
Description: Acute rejections[1] between initiation of sirolimus withdrawal and end of study
  1] Acute rejection is defined as a biopsy-proven rejection: a renal biopsy demonstrates acute cellular or humoral rejection of Banff[2] Grade 1B or greater; or presumed rejection in the absence of biopsy-proven rejection, the participant is treated for an unexplained 20% increase in serum creatinine.
  [2] Reference: Racusen LC, Solez K, Colvin RB et al,The Banff 97 working classification of renal allograft pathology. Kidney Int,55: 713-723, 1999
Time Frame: Initiation of sirolimus to end of study (up to four years post-transplant)
Population: Sirolimus withdrawal initiation participant sample
Measure: Number; unit: Rejection Events
Arm/Group | Alemtuzumab
Number analyzed (Participants) | 2
Rejection Events | 0
Statistical Analysis 1: Comparison: Alemtuzumab; Test type: Superiority or Other; 95% Confidence Interval; Exact Binomial; Proportion with acute rejection = 0, 95% CI 2-sided [0.0 to 0.7]

4. Secondary Outcome: Time From Transplantation to Acute Rejection in Participants for Whom Sirolimus Withdrawal Was Not Initiated
Description: Time (days) to acute rejection[1] for participants where sirolimus was not initiated
  1] Acute rejection is defined as a biopsy-proven rejection: a renal biopsy demonstrates acute cellular or humoral rejection of Banff[2] Grade 1B or greater; or presumed rejection in the absence of biopsy-proven rejection, the participant is treated for an unexplained 20% increase in serum creatinine.
  [2] Reference: Racusen LC, Solez K, Colvin RB et al,The Banff 97 working classification of renal allograft pathology. Kidney Int,55: 713-723, 1999
Time Frame: Transplantation to acute rejection (up to four years post-transplantation)
Population: Participants for whom sirolimus withdrawal was not initiated
Measure: Number; unit: Days
Arm/Group | Alemtuzumab
Number analyzed (Participants) | 1
Days | 274

5. Secondary Outcome: Time From Transplantation to Acute Rejection in Participants for Whom Acute Rejection Occurred During the 1 Year Post-transplant Period
Description: Time (days) to acute rejection[1] for participants occurring during the year following transplantation
  1] Acute rejection is defined as a biopsy-proven rejection: a renal biopsy demonstrates acute cellular or humoral rejection of Banff[2] Grade 1B or greater; or presumed rejection in the absence of biopsy-proven rejection, the participant is treated for an unexplained 20% increase in serum creatinine.
  [2] Reference: Racusen LC, Solez K, Colvin RB et al,The Banff 97 working classification of renal allograft pathology. Kidney Int,55: 713-723, 1999
Time Frame: Transplantation to acute rejection (up to one year post-transplant)
Population: Participants with acute rejections for whom sirolimus withdrawal was not initiated
Measure: Number; unit: Days
Arm/Group | Alemtuzumab
Number analyzed (Participants) | 1
Days | 274

6. Secondary Outcome: Number of Deaths Stratified by Sirolimus Withdrawal Status
Description: Participants who died during the study, all cause(s)
Time Frame: Transplantation to Death (up to four years post-transplant)
Population: Intent-to-treat
Measure: Number; unit: deaths
Groups:
- Alemtuzumab (Withdrawn From Sirolimus): Recipients of first kidney transplants (0-3 HLA antigen mismatch) received induction therapy with alemtuzumab (1 dose [30 mg]each day, Days 0 [transplant day], 1 and 2, administered intravenously) , tacrolimus (the dose was initially 2 mg twice daily by mouth, and adjusted to maintain target blood levels of 4 to 8 ng/mL from Day 1 to Day 60) and sirolimus (the initial dose was 2 mg/day by mouth started <= 48 hours post-transplant, subsequently adjusted to achieve trough levels of 8 to 12 ng/mL through Month 12), followed by sirolimus withdrawal as tolerated
- Alemtuzumab (Not Withdrawn From Sirolimus): Recipients of first kidney transplants (0-3 HLA antigen mismatch) received induction therapy with alemtuzumab (1 dose [30 mg]each day, Days 0 [transplant day], 1 and 2, administered intravenously) , tacrolimus (the dose was initially 2 mg twice daily by mouth, and adjusted to maintain target blood levels of 4 to 8 ng/mL from Day 1 to Day 60) and sirolimus (the initial dose was 2 mg/day by mouth started <= 48 hours post-transplant, subsequently adjusted to achieve trough levels of 8 to 12 ng/mL through Month 12)
Arm/Group | Alemtuzumab (Withdrawn From Sirolimus) | Alemtuzumab (Not Withdrawn From Sirolimus)
Number analyzed (Participants) | 2 | 8
deaths | 0 | 0
Statistical Analysis 1: Comparison: Alemtuzumab (Withdrawn From Sirolimus) vs Alemtuzumab (Not Withdrawn From Sirolimus); Test type: Superiority or Other; 95% Confidence Interval; Exact Binomial; Exact Binomial = 0, 95% CI 2-sided [0.0 to 0.3]

7. Secondary Outcome: Number of Participants Who Experienced Graft Loss Stratified by Sirolimus Withdrawal Status
Description: Participants who experienced graft loss[1] during study
  [1]Graft loss is defined as the institution of chronic dialysis (at least 6 consecutive weeks, excluding participants with delayed graft function), transplant nephrectomy, or retransplantation
Time Frame: Transplantation to Graft Loss (up to four years post-transplantation)
Population: Intent-to-treat
Measure: Number; unit: participants
Arm/Group | Alemtuzumab (Withdrawn From Sirolimus) | Alemtuzumab (Not Withdrawn From Sirolimus)
Number analyzed (Participants) | 2 | 8
participants | 0 | 0
Statistical Analysis 1: Comparison: Alemtuzumab (Withdrawn From Sirolimus) vs Alemtuzumab (Not Withdrawn From Sirolimus); Test type: Superiority or Other; 95% Confidence Interval; Exact Binomial for all participants (n=10); Exact Binomial = 0, 95% CI 2-sided [0.0 to 0.3]

8. Secondary Outcome: Number of Severe Acute Rejections Stratified by Sirolimus Withdrawal Status
Description: Participants who experienced severe acute rejections[1] during study
  1. Severe acute rejection is defined as that which requires treatment with anti-lymphocyte antibody or is histologically evaluated as Type IIA or greater using the Banff 1997 criteria[2]
  2. Reference: Racusen LC, Solez K, Colvin RB et al,The Banff 97 working classification of renal allograft pathology. Kidney Int,55: 713-723, 1999
Time Frame: Transplantation to severe acute rejection (up to four years post-transplantation)
Population: Intent-to-treat
Measure: Number; unit: Rejection Events
Arm/Group | Alemtuzumab (Withdrawn From Sirolimus) | Alemtuzumab (Not Withdrawn From Sirolimus)
Number analyzed (Participants) | 2 | 8
Rejection Events | 0 | 0
Statistical Analysis 1: Comparison: Alemtuzumab (Withdrawn From Sirolimus); Test type: Superiority or Other; 95% Confidence Interval; Exact Binomial for Not Withdrawn Group; Exact Binomial = 0, 95% CI 2-sided [0.0 to 0.4]
Statistical Analysis 2: Comparison: Alemtuzumab (Not Withdrawn From Sirolimus); Test type: Superiority or Other; 95% Confidence Interval; Exact Binomial for Withdrawn Group; Exact Binomial = 0, 95% CI 2-sided [0.0 to 0.8]

9. Secondary Outcome: Number of Participants Requiring Anti-lymphocyte Therapy for an Acute Rejection, Stratified by Sirolimus Withdrawal Status
Description: Participants who experienced acute rejection[1] during study which required anti-lymphocyte (OKT3, ATG) therapy
  1] Acute rejection is defined as a biopsy-prove rejection: a renal biopsy demonstrates acute cellular or humoral rejection of Banff[2] Grade 1B or greater; or presumed rejection in the absence of biopsy-proven rejection, the participant is treated for an unexplained 20% increase in serum creatinine.
  [2] Reference: Racusen LC, Solez K, Colvin RB et al,The Banff 97 working classification of renal allograft pathology. Kidney Int,55: 713-723, 1999
Time Frame: Transplantation to acute rejection (up to four years post-transplantation)
Population: Intent-to-treat
Measure: Number; unit: participants
Arm/Group | Alemtuzumab (Withdrawn From Sirolimus) | Alemtuzumab (Not Withdrawn From Sirolimus)
Number analyzed (Participants) | 2 | 8
participants | 0 | 0
Statistical Analysis 1: Comparison: Alemtuzumab (Withdrawn From Sirolimus); Test type: Superiority or Other; 95% Confidence Interval; Exact Binomial for Not Withdrawn Group; Exact Binomial = 0, 95% CI 2-sided [0.0 to 0.4]
Statistical Analysis 2: Comparison: Alemtuzumab (Not Withdrawn From Sirolimus); Test type: Superiority or Other; 95% Confidence Interval; Exact Binomial for Withdrawn Group; Exact Binomial = 0, 95% CI 2-sided [0.0 to 0.8]

10. Secondary Outcome: Number of Alemtuzumab Associated Adverse Events, Stratified by Sirolimus Withdrawal Status
Time Frame: Transplantation to end of study (up to four years post-transplant)
Population: Intent-to-treat
Measure: Number; unit: adverse events
Arm/Group | Alemtuzumab (Withdrawn From Sirolimus) | Alemtuzumab (Not Withdrawn From Sirolimus)
Number analyzed (Participants) | 2 | 8
adverse events | 2 | 8

11. Secondary Outcome: Number of Tacrolimus Associated Adverse Events, Stratified by Sirolimus Withdrawal Status
Time Frame: Transplantation to end of study (up to four years post-transplant)
Population: Intent-to-treat
Measure: Number; unit: adverse events
Arm/Group | Alemtuzumab (Withdrawn From Sirolimus) | Alemtuzumab (Not Withdrawn From Sirolimus)
Number analyzed (Participants) | 2 | 8
adverse events | 0 | 2

12. Secondary Outcome: Number of Sirolimus Associated Adverse Events, Stratified by Sirolimus Withdrawal Status
Time Frame: Transplantation to end of study (up to four years post-transplant)
Population: Intent-to-treat
Measure: Number; unit: adverse events
Arm/Group | Alemtuzumab (Withdrawn From Sirolimus) | Alemtuzumab (Not Withdrawn From Sirolimus)
Number analyzed (Participants) | 2 | 8
adverse events | 2 | 7

13. Secondary Outcome: Number of Side Effects of Conventional Immunosuppression, Stratified by Withdrawal Status
Description: Side effects of conventional immunosuppression include increased body weight and hypertension
Time Frame: Transplantation to end of study (up to four years post-transplant)
Population: Intent-to-treat
Measure: Number; unit: side effects
Arm/Group | Alemtuzumab (Withdrawn From Sirolimus) | Alemtuzumab (Not Withdrawn From Sirolimus)
Number analyzed (Participants) | 2 | 8
side effects | 2 | 6

14. Secondary Outcome: Change in Renal Function as Measured by Serum Creatinine, Stratified by Withdrawal Status
Description: Mean change from transplantation to Month 48 in serum creatinine. Normal serum creatinine range is from 0.7 - 1.4 mg/dL. In a transplant population, starting serum creatinine is higher than normal range. A negative change indicates better renal function
Time Frame: Transplantation to end of study (up to four years post-transplant)
Population: Intent-to-treat
Measure: Mean (Standard Deviation); unit: mg/dL
Arm/Group | Alemtuzumab (Withdrawn From Sirolimus) | Alemtuzumab (Not Withdrawn From Sirolimus)
Number analyzed (Participants) | 2 | 8
mg/dL | -4.2 (2.3) | -5.4 (2.7)

ADVERSE EVENTS:
Arm/Group | Alemtuzumab
Serious Adverse Events (participants affected / at risk) | 5/10
Other Adverse Events (participants affected / at risk) | 10/10
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Alemtuzumab (N=10)
Anaemia (Blood and lymphatic system disorders) | 1 (1)
Ileus (Gastrointestinal disorders) | 1 (1)
Transplant rejection (Immune system disorders) | 1 (1)
Escherichia sepsis (Infections and infestations) | 1 (1)
Gas gangrene (Infections and infestations) | 1 (1)
Pneumonia klebsiella (Infections and infestations) | 1 (1)
Incisional hernia (Injury, poisoning and procedural complications) | 1 (1)
Osteonecrosis (Musculoskeletal and connective tissue disorders) | 1 (2)
Renal cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1)
Syncope (Nervous system disorders) | 1 (1)
Proteinuria (Renal and urinary disorders) | 1 (1)
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Deep vein thrombosis (Vascular disorders) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Alemtuzumab (N=10)
Anaemia (Blood and lymphatic system disorders) | 8 (17)
Leukocytosis (Blood and lymphatic system disorders) | 2 (2)
Leukopenia (Blood and lymphatic system disorders) | 8 (14)
Lymphadenitis (Blood and lymphatic system disorders) | 1 (1)
Lymphadenopathy (Blood and lymphatic system disorders) | 1 (1)
Lymphopenia (Blood and lymphatic system disorders) | 10 (10)
Neutropenia (Blood and lymphatic system disorders) | 3 (4)
Thrombocytopenia (Blood and lymphatic system disorders) | 3 (3)
Atrial fibrillation (Cardiac disorders) | 1 (2)
Pericardial effusion (Cardiac disorders) | 1 (1)
Sinus tachycardia (Cardiac disorders) | 5 (6)
Supraventricular extrasystoles (Cardiac disorders) | 1 (1)
Tachycardia (Cardiac disorders) | 1 (1)
Ventricular extrasystoles (Cardiac disorders) | 1 (1)
Cushingoid (Endocrine disorders) | 1 (1)
Hyperparathyroidism (Endocrine disorders) | 1 (1)
Hyperparathyroidism secondary (Endocrine disorders) | 1 (1)
Hyperthyroidism (Endocrine disorders) | 1 (3)
Abnormal sensation in eye (Eye disorders) | 1 (1)
Blepharospasm (Eye disorders) | 1 (1)
Cataract (Eye disorders) | 1 (1)
Conjunctivitis (Eye disorders) | 1 (1)
Eyelid oedema (Eye disorders) | 1 (1)
Vision blurred (Eye disorders) | 2 (2)
Visual acuity reduced (Eye disorders) | 2 (2)
Abdominal discomfort (Gastrointestinal disorders) | 1 (1)
Abdominal distension (Gastrointestinal disorders) | 6 (6)
Abdominal hernia (Gastrointestinal disorders) | 1 (1)
Abdominal pain (Gastrointestinal disorders) | 3 (3)
Abdominal pain lower (Gastrointestinal disorders) | 1 (1)
Aphthous stomatitis (Gastrointestinal disorders) | 2 (2)
Constipation (Gastrointestinal disorders) | 5 (7)
Diarrhoea (Gastrointestinal disorders) | 6 (14)
Dry mouth (Gastrointestinal disorders) | 1 (1)
Eructation (Gastrointestinal disorders) | 1 (1)
Flatulence (Gastrointestinal disorders) | 2 (2)
Gastrointestinal sounds abnormal (Gastrointestinal disorders) | 7 (7)
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 2 (2)
Glossodynia (Gastrointestinal disorders) | 1 (1)
Ileus (Gastrointestinal disorders) | 2 (2)
Localised intraabdominal fluid collection (Gastrointestinal disorders) | 1 (1)
Mouth ulceration (Gastrointestinal disorders) | 2 (2)
Nausea (Gastrointestinal disorders) | 6 (10)
Sensitivity of teeth (Gastrointestinal disorders) | 1 (1)
Stomatitis (Gastrointestinal disorders) | 1 (1)
Toothache (Gastrointestinal disorders) | 2 (2)
Vomiting (Gastrointestinal disorders) | 3 (5)
Chills (General disorders) | 1 (1)
Fatigue (General disorders) | 5 (7)
Gait disturbance (General disorders) | 1 (1)
Generalised oedema (General disorders) | 5 (6)
Infusion site extravasation (General disorders) | 1 (1)
Malaise (General disorders) | 2 (2)
Oedema (General disorders) | 2 (2)
Oedema peripheral (General disorders) | 9 (19)
Pain (General disorders) | 1 (1)
Pyrexia (General disorders) | 6 (11)
Xerosis (General disorders) | 1 (1)
Gallbladder polyp (Hepatobiliary disorders) | 1 (1)
Hepatic cyst (Hepatobiliary disorders) | 1 (1)
Hypersensitivity (Immune system disorders) | 1 (1)
Seasonal allergy (Immune system disorders) | 3 (5)
Bronchitis (Infections and infestations) | 1 (1)
Cellulitis (Infections and infestations) | 2 (2)
Chromoblastomycosis (Infections and infestations) | 1 (1)
Cytomegalovirus viraemia (Infections and infestations) | 2 (2)
Escherichia urinary tract infection (Infections and infestations) | 1 (1)
Eyelid folliculitis (Infections and infestations) | 1 (1)
Folliculitis (Infections and infestations) | 1 (2)
Gastroenteritis viral (Infections and infestations) | 3 (5)
Herpes zoster (Infections and infestations) | 1 (1)
Human polyomavirus infection (Infections and infestations) | 1 (1)
Incision site cellulitis (Infections and infestations) | 1 (1)
Influenza (Infections and infestations) | 1 (1)
Klebsiella infection (Infections and infestations) | 2 (3)
Nasopharyngitis (Infections and infestations) | 1 (1)
Oral candidiasis (Infections and infestations) | 1 (1)
Oral herpes (Infections and infestations) | 1 (1)
Pharyngitis (Infections and infestations) | 1 (1)
Pneumonia cryptococcal (Infections and infestations) | 1 (1)
Sinusitis (Infections and infestations) | 4 (9)
Upper respiratory tract infection (Infections and infestations) | 5 (8)
Urinary tract infection (Infections and infestations) | 2 (4)
Urinary tract infection bacterial (Infections and infestations) | 2 (3)
Urinary tract infection staphylococcal (Infections and infestations) | 1 (2)
Viral upper respiratory tract infection (Infections and infestations) | 1 (1)
Back injury (Injury, poisoning and procedural complications) | 1 (1)
Chronic allograft nephropathy (Injury, poisoning and procedural complications) | 2 (2)
Complications of transplanted kidney (Injury, poisoning and procedural complications) | 1 (1)
Contusion (Injury, poisoning and procedural complications) | 3 (3)
Dialysis device complication (Injury, poisoning and procedural complications) | 1 (1)
Drug toxicity (Injury, poisoning and procedural complications) | 1 (1)
Excoriation (Injury, poisoning and procedural complications) | 1 (1)
Fall (Injury, poisoning and procedural complications) | 1 (1)
Incision site complication (Injury, poisoning and procedural complications) | 10 (12)
Incision site pain (Injury, poisoning and procedural complications) | 10 (12)
Incisional hernia (Injury, poisoning and procedural complications) | 1 (1)
Incorrect dose administered (Injury, poisoning and procedural complications) | 1 (1)
Open wound (Injury, poisoning and procedural complications) | 1 (1)
Perinephric collection (Injury, poisoning and procedural complications) | 1 (1)
Post procedural haematoma (Injury, poisoning and procedural complications) | 1 (1)
Renal injury (Injury, poisoning and procedural complications) | 1 (1)
Seroma (Injury, poisoning and procedural complications) | 1 (1)
Skin laceration (Injury, poisoning and procedural complications) | 1 (1)
Alanine aminotransferase increased (Investigations) | 6 (6)
Aspartate aminotransferase increased (Investigations) | 3 (3)
Blood alkaline phosphatase increased (Investigations) | 5 (7)
Blood creatinine increased (Investigations) | 4 (6)
Blood lactate dehydrogenase increased (Investigations) | 6 (7)
Breath sounds abnormal (Investigations) | 10 (12)
Gamma-glutamyltransferase increased (Investigations) | 4 (6)
Oxygen saturation decreased (Investigations) | 1 (1)
Urine output decreased (Investigations) | 1 (1)
Weight decreased (Investigations) | 1 (1)
Weight increased (Investigations) | 6 (8)
Dehydration (Metabolism and nutrition disorders) | 4 (4)
Dyslipidaemia (Metabolism and nutrition disorders) | 3 (3)
Gout (Metabolism and nutrition disorders) | 1 (1)
Hypercalcaemia (Metabolism and nutrition disorders) | 1 (1)
Hyperglycaemia (Metabolism and nutrition disorders) | 3 (3)
Hyperkalaemia (Metabolism and nutrition disorders) | 1 (1)
Hyperlipidaemia (Metabolism and nutrition disorders) | 9 (11)
Hypertriglyceridaemia (Metabolism and nutrition disorders) | 3 (3)
Hypocalcaemia (Metabolism and nutrition disorders) | 1 (1)
Hypokalaemia (Metabolism and nutrition disorders) | 2 (3)
Hypomagnesaemia (Metabolism and nutrition disorders) | 3 (3)
Hyponatraemia (Metabolism and nutrition disorders) | 2 (3)
Hypophosphataemia (Metabolism and nutrition disorders) | 6 (7)
Increased appetite (Metabolism and nutrition disorders) | 1 (1)
Metabolic acidosis (Metabolism and nutrition disorders) | 2 (3)
Obesity (Metabolism and nutrition disorders) | 2 (2)
Vitamin D deficiency (Metabolism and nutrition disorders) | 3 (3)
Arthralgia (Musculoskeletal and connective tissue disorders) | 3 (4)
Back pain (Musculoskeletal and connective tissue disorders) | 2 (2)
Joint stiffness (Musculoskeletal and connective tissue disorders) | 1 (1)
Muscle spasms (Musculoskeletal and connective tissue disorders) | 1 (1)
Muscle twitching (Musculoskeletal and connective tissue disorders) | 1 (1)
Muscular weakness (Musculoskeletal and connective tissue disorders) | 1 (1)
Musculoskeletal chest pain (Musculoskeletal and connective tissue disorders) | 1 (1)
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 1 (1)
Myalgia (Musculoskeletal and connective tissue disorders) | 5 (6)
Neck pain (Musculoskeletal and connective tissue disorders) | 1 (1)
Osteopenia (Musculoskeletal and connective tissue disorders) | 4 (4)
Osteoporosis (Musculoskeletal and connective tissue disorders) | 1 (1)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 4 (6)
Pain in jaw (Musculoskeletal and connective tissue disorders) | 1 (1)
Plantar fasciitis (Musculoskeletal and connective tissue disorders) | 1 (1)
Lung neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1)
Burning sensation (Nervous system disorders) | 1 (1)
Dizziness (Nervous system disorders) | 3 (3)
Dysgeusia (Nervous system disorders) | 1 (1)
Headache (Nervous system disorders) | 3 (6)
Hypoaesthesia (Nervous system disorders) | 1 (1)
Neuropathy peripheral (Nervous system disorders) | 3 (3)
Restless legs syndrome (Nervous system disorders) | 1 (1)
Tremor (Nervous system disorders) | 2 (2)
Agitation (Psychiatric disorders) | 1 (1)
Disorientation (Psychiatric disorders) | 1 (1)
Dysuria (Renal and urinary disorders) | 1 (1)
Haematuria (Renal and urinary disorders) | 6 (6)
Hydronephrosis (Renal and urinary disorders) | 1 (1)
Hydroureter (Renal and urinary disorders) | 1 (1)
Micturition urgency (Renal and urinary disorders) | 1 (1)
Nephropathy toxic (Renal and urinary disorders) | 3 (3)
Pollakiuria (Renal and urinary disorders) | 1 (2)
Proteinuria (Renal and urinary disorders) | 4 (6)
Pyelocaliectasis (Renal and urinary disorders) | 2 (2)
Renal infarct (Renal and urinary disorders) | 1 (1)
Ureteral disorder (Renal and urinary disorders) | 1 (1)
Urethral stenosis (Renal and urinary disorders) | 1 (1)
Urinary retention (Renal and urinary disorders) | 1 (1)
Ovarian cyst (Reproductive system and breast disorders) | 1 (1)
Apnoea (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Atelectasis (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Cough (Respiratory, thoracic and mediastinal disorders) | 3 (4)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 4 (5)
Dyspnoea exertional (Respiratory, thoracic and mediastinal disorders) | 2 (3)
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Productive cough (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Pulmonary congestion (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Pulmonary oedema (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Rhinorrhoea (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Wheezing (Respiratory, thoracic and mediastinal disorders) | 2 (2)
Acne (Skin and subcutaneous tissue disorders) | 2 (4)
Actinic keratosis (Skin and subcutaneous tissue disorders) | 1 (1)
Blister (Skin and subcutaneous tissue disorders) | 1 (1)
Dermatitis (Skin and subcutaneous tissue disorders) | 1 (1)
Erythema (Skin and subcutaneous tissue disorders) | 1 (1)
Ingrown hair (Skin and subcutaneous tissue disorders) | 1 (1)
Nail discolouration (Skin and subcutaneous tissue disorders) | 1 (1)
Pain of skin (Skin and subcutaneous tissue disorders) | 1 (1)
Pruritus (Skin and subcutaneous tissue disorders) | 10 (11)
Rash (Skin and subcutaneous tissue disorders) | 5 (5)
Urticaria (Skin and subcutaneous tissue disorders) | 6 (6)
Deep vein thrombosis (Vascular disorders) | 1 (1)
Flushing (Vascular disorders) | 2 (2)
Haematoma (Vascular disorders) | 1 (1)
Hypertension (Vascular disorders) | 6 (10)
Hypotension (Vascular disorders) | 4 (4)
Lymphocele (Vascular disorders) | 1 (1)

LIMITATIONS AND CAVEATS:
The absence of a control group in this pilot trial precludes any comparison between alemtuzumab-induced patients with further minimization and patients with more conventional immunosuppressive approaches, and is a limitation of the current study

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No